CLINICAL TRIAL: NCT05450484
Title: Optical PD-L1 Imaging Using Quantitative Fluorescence Endoscopy in Locally Advanced Esophageal Cancer Using Durvalumab-680LT: a Multicenter Feasibility and Safety Study
Brief Title: Quantitative Fluorescence Endoscopy Using Durvalumab-680LT in Esophageal Cancer
Acronym: OPTIC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202000424
Record Dates: First submitted 2022-06-13; First posted 2022-07-08 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab-680LT (Experimental)
  Interventions: Drug: Fluorescence endoscopy using durvalumab-680LT

INTERVENTIONS:
Drug: Fluorescence endoscopy using durvalumab-680LT — Tracer administration: The PD-L1-targeted fluorescent tracer durvalumab-680LT will be administered intravenously 2-4 days prior to the endoscopy at the UMCG. Afterwards, patients will be monitored for half an hour by measurements of vital parameters for potential side-effects, such as infusion-related reactions.
  Endoscopy procedure: Patients will undergo two endoscopies, before and after neoadjuvant therapy. First, routine high-definition white-light (HD-WL) inspection is used. Quantification of fluorescence using multi-diameter single fiber reflectance/single fiber fluorescence (MDSFR/SFF) spectroscopy will be performed both in vivo and ex vivo. Subsequently, fluorescence molecular endoscopy (FME) and endoscopic ultrasound (EUS) will be performed. EUS enables single fiber reflectance/single fiber fluorescence (SFR/SFF) spectroscopy measurements via fine needle aspiration (FNA) to gain insight in the drug distribution throughout the tumor. Additionally, biopsies will be obtained.

SUMMARY:
Treatment of patients with locally advanced esophageal cancer (EC) is multidisciplinary and consists of neoadjuvant therapy followed by surgical removal of the esophageal tumor and potentially tumor positive lymph nodes. The beneficial effect of the addition of immunotherapy to improve response rates to current treatment strategies has been investigated response to, since only 16 to 43% of EC patients achieve a pathological complete response (pCR) after neoadjuvant therapy and a pCR is associated with better long-term outcomes. Unfortunately, not all patients respond to immunotherapy and the knowledge about biomarkers that predict response to therapy are required. A promising novel parameter is tumor programmed death-ligand 1 (PD-L1) expression, one of the immune checkpoints targeted by cancer immunotherapy. Studies performed in patients with various solid tumors demonstrate improved response to immunotherapy and survival benefit in patients with higher PD-L1 expression. Nonetheless, not all patients with high PD-L1 expression show benefit and some without expression do. Moreover, mostly biopsy-based tests are used to assess PD-L1 status, although these tests are prone to errors, partly due to heterogeneity in tissue expression. Novel methods are needed to gain more insight in the PD-L1 expression in order to better select patients who are likely to benefit from immunotherapy. The investigators hypothesize that quantitative fluorescence endoscopy using the tracer durvalumab-680LT targeting PD-L1 is a promising technique to investigate the heterogeneity of PD-L1 expression.

ELIGIBILITY:
Inclusion Criteria:

* Lesion suspected for locally advanced EC (cT1b-4a N0-3 M0)
* Indication for neoadjuvant therapy
* Age ≥ 18 years;
* Written informed consent.

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent according to treating medical physician;
* Concurrent uncontrolled medical conditions according to treating medical physician;
* Medical history of auto-immune disease
* Pregnancy or breast feeding. A negative pregnancy test must be available for women of childbearing potential (i.e. premenopausal women with intact reproductive organs and women less than two years after menopause);
* Irradical endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of the primary tumor prior to start of neoadjuvant therapy according to the patient's medical history;
* Received an investigational drug within 30 days prior to the dose of durvalumab-680LT according to the patient's medical history;
* History of infusion reactions to durvalumab or other monoclonal antibodies according to the patient's medical history;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
1) Evaluating the heterogeneity of the PD-L1 tumor expression before and after neoadjuvant therapy using quantitative fluorescence endoscopy using the PD-L1-targeted fluorescent tracer durvalumab-680LT | Within 12 months after the study procedures
  Quantification of the fluorescent durvalumab-680LT signal, both in vivo and ex vivo, using our spectroscopy device before and after neoadjudant treatment.
2) Incidence of (severe) adverse events (SAE/AEs) related to administration of durvalumab-680LT assessed by CTCAE | Up to one week after tracer administration
  Safety of durvalumab-680LT administration will be assessed by using Common Terminology Criteria for Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No